CLINICAL TRIAL: NCT07032545
Title: Metabotyping of a Functional Food, Broccoli Microgreen, in Obese Breast Cancer Survivors
Brief Title: Metabotyping of Broccoli Microgreen in Obese Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Yuanyuan (Rose) Li, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00113949
Record Dates: First submitted 2025-06-10; First posted 2025-06-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity and Overweight; Breast Cancer Survivorship
Keywords: breast cancer; broccoli microgreen; obesity; survivorship; gut microbiome; metabolomics; metabotyping
MeSH Terms: conditions — Obesity; Overweight; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single arm pilot intervention trial and all participants will be asked to consume allocated broccoli microgreen for 2 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMG (Experimental): All participants are in BMG group and will consume one serving size (one cup, ~57 gram) of raw BMG daily for 2-week period of time.
  Interventions: Other: Broccoli microgreen (BMG)

INTERVENTIONS:
Other: Broccoli microgreen (BMG) — All participants will consume one serving size (one cup, ~57 gram) of raw BMG daily for 2-week period of time.

SUMMARY:
Obesity can pose significant challenges to maintaining long-term health in cancer survivors by increasing their risk of cancer coming back. Eating a healthy diet is an important way to help manage weight and improve overall health. Broccoli microgreens (BMG) are young broccoli plants packed with nutrients, and research suggests they may help prevent cancer.

Previous studies in mice showed that BMG can improve gut health and metabolism, leading to better health outcomes in obese animals. This study will test whether BMG can be a useful addition to the diet of obese breast cancer (BC) survivors who have a higher risk of their cancer returning.

24 obese BC survivors will be invited to eat one serving (one cup, ~57 gram) of fresh BMG every day for two weeks. This will help understand if people can stick to this diet, how their bodies respond, and whether it affects metabolism and inflammation-two key factors linked to cancer risk. Biological markers such as body fat, glucose and lipids as well as gut bacterial changes will be analyzed to see how BMG affects individual health.

This study may help create new diet strategies to improve health, reduce cancer risk, and support long-term recovery in cancer patients who are overweight or obese. In the future, this research could help doctors personalize nutrition plans to better support cancer survivors.

DETAILED DESCRIPTION:
In this pilot clinical trial, 24 obese BC survivors from the University of Maryland Medical Center in Baltimore will be recruited to participate in a single-arm 2-week BMG (broccoli microgreen) intervention trial. Several outcomes will be tested, including study feasibility, patient compliance of one serving size of raw BMG and metabolic parameter changes. Biological samples such as blood and fecal samples as well as study questionnaires will be collected at baseline and 2 weeks post-intervention to measure the outcomes. The main hypothesis of this study is that incorporating the proposed BMG quantity into daily meals is feasible in obese BC survivors. The secondary hypothesis is that BMG may improve the metabolic profiles and gut health in obese subjects. This proof-of-concept prospective study will provide important clinical insights into beneficial effects of BMG on mitigating obesity and related metabolic disorders, which strategies may complement traditional survivorship management and support long-term health outcomes for BC survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Had a diagnosis of breast cancer (Stage I-III)
* 2 to 60 months post-curative treatment (surgery, chemotherapy, and/or radiation)
* BMI > 30 kg/m² (obese classification)
* Willing to avoid cruciferous vegetables during the study
* Able to sign an IRB-approved consent form

Exclusion Criteria:

* Have any contraindications to the proposed nutrition intervention as identified by their medical provider, their designee, or the study team (e.g., GI conditions, medication requirements, pregnancy, breastfeeding, recent history of an eating disorder).
* Allergy or intolerance to cruciferous vegetables
* Currently taking broccoli extract supplements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as Assessed by the Percentage of Participants Who Enrolled and Completed the Study | 14 days
  Feasibility will be assessed by calculating the percentage of participants who enrolled and completed the study by providing evaluable data at baseline, during the BMG intervention and after 2-weeks treatment.
Compliance, as Assessed by the Percentage of the Participants Who Adhere to the Assigned BMG Intervention | 14 days
  Compliance will be assessed by measuring the percent of the participants who consume the assigned BMG through the recommended cooking method during the 2-weeks of intervention period.

SECONDARY OUTCOMES:
Body Composition, as Assessed by the Percentage of the Body Fat | 14 days
  Body fat composition will be determined by measuring the percentage of body fat by a Handheld Body Composition Monitor. Data will be analyzed by comparing the mean change before and after the BMG dietary treatment using paired samples t-tests. Statistical significance will be assumed at p < 0.05, and results will be based on two-tailed statistical tests.
Blood Glucose, as Assessed by Fasting Blood Glucose Level | 14 days
  The fasting blood glucose level will be measured to determine the glucose concentration changes before and after the BMG dietary treatment. Data will be analyzed by comparing the mean change of the fasting glucose concentrations before and after the BMG dietary treatment using paired samples t-tests. Statistical significance will be assumed at p < 0.05, and results will be based on two-tailed statistical tests.
Blood Lipids, as Assessed by Blood Lipid Concentrations | 14 days
  The blood lipids including total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides will be measured to determine the lipid concentration changes before and after the BMG dietary treatment. Data will be analyzed by comparing the mean change of the individual lipid concentrations before and after the intervention using paired samples t-tests. Statistical significance will be assumed at p < 0.05, and results will be based on two-tailed statistical tests.
The Gut microbiome, as Assessed by the Bacterial Composition Changes | 14 days
  Gut microbial composition changes will be evaluated by sequencing-based methods before and after the BMG diet intervention. Key parameters for assessing microbiome changes include alpha and beta diversity changes as well as the individual bacterial composition differences in response to BMG intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan (Rose) Li, M.D., Ph.D., Principal Investigator — University of Maryland
Locations (1):
- Breast Evaluation and Treatment Program, University of Maryland Marlene and Stewart Greenebaum Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bankole T, Ma T, Arora I, Lei Z, Raju M, Li Z, Li Y. The Effect of Broccoli Glucoraphanin Supplementation on Ameliorating High-Fat-Diet-Induced Obesity through the Gut Microbiome and Metabolome Interface. Mol Nutr Food Res. 2024 May;68(9):e2300856. doi: 10.1002/mnfr.202300856. Epub 2024 Apr 27. PMID 38676466
- [Background] Turner ER, Luo Y, Buchanan RL. Microgreen nutrition, food safety, and shelf life: A review. J Food Sci. 2020 Apr;85(4):870-882. doi: 10.1111/1750-3841.15049. Epub 2020 Mar 6. PMID 32144769
- [Background] Wojdylo A, Nowicka P, Tkacz K, Turkiewicz IP. Sprouts vs. Microgreens as Novel Functional Foods: Variation of Nutritional and Phytochemical Profiles and Their In Vitro Bioactive Properties. Molecules. 2020 Oct 12;25(20):4648. doi: 10.3390/molecules25204648. PMID 33053861